CLINICAL TRIAL: NCT04470115
Title: Femoral Nerve Block Together With Lateral Femoral Cutaneous Nerve Block and Sedation as Anesthesia Among High Risk Patients With Intertrochanteric Fracture Repair Surgery
Brief Title: Blocks for Intertrochanteric Fracture Repair Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Jakub Klimkiewicz, Principal Investigator, Military Institute od Medicine National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01_2019
Record Dates: First submitted 2020-07-01; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Intertrochanteric Fractures
Keywords: intratrochanteric fracture; general anesthesia; femoral nerve block; lateral femoral cutaneous nerve block
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator): Patients will receive general endotracheal anesthesia with propofol, fentanyl, sevoflurane and rocuronium.
  Interventions: Other: General anesthesia
- Regional anesthesia (Experimental): Patients will receive femoral and lateral femoral cutaneous nerves block under ultrasonographical guidance before operation.During surgical procedure they will receive deep sedation with propofol.
  Interventions: Other: Regional anesthesia- femoral and lateral femoral cutaneous nerve blocks

INTERVENTIONS:
Other: General anesthesia — Patients will receive general endotracheal anesthesia with typical drugs used (propofol, fentanyl, sevoflurane). the exact dose of the drug will be on the discretion of anesthesia provider, according to good clinical practice.
  Arms: General anesthesia
Other: Regional anesthesia- femoral and lateral femoral cutaneous nerve blocks — The femoral nerve (FN) is identified with ultrasound. The needle is inserted in-plane, from lateral to medial. We administer 15 to 17ml of local anesthetic (0.5 to 0.75% ropivacaine). After good anesthetic spread on FN we identify lateral femoral cutaneous nerve (LFCN) in its expected location 2-3 cm below inguinal ligament, laterally to sartorius muscle and inject usually 4 to 5 ml of local anesthetic. Oxygen 2-3 l/min is given via face mask to maintain Sp02 and the block is followed by sedation. Sedation is achieved with boluses of propofol to enable procedure and maintain patient in comfort. We aim to keep the depth of sedation at Ramsay sedation scale of 4. Whether it is possible we use loud verbal stimulus, if it is not we use gently glabella tap to assess depth of sedation. Patient is breathing spontaneously during the whole surgery. After surgical field is prepared, surgeon infiltrates expected entry points of intramedullary nail system with 0,5% lidocaine.
  Arms: Regional anesthesia

SUMMARY:
This single-center open label study compares the outcomes of surgical repair of intratrochanteric fracture under general anesthetic or peripheral nerve blocks.

DETAILED DESCRIPTION:
This single-center open label study compares the outcomes of surgical repair of intratrochanteric fracture under general anesthetic or peripheral nerve blocks.

Patients are high risk individuals scheduled for intratrochanteric fracture repair, with contraindications to spinal anesthesia. One group will receive general endotracheal anesthetic, the other femoral and lateral femoral cutaneous nerve with deep sedation.

Mortality, morbidity (major cardiovascular incidents,delirium, pneumonia), pain scores and opioid consumption will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* intratrochanteric fracture
* need for surgery
* contraindications for spinal anesthesia

Exclusion Criteria:

* allergy to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients surviving 30 days after the surgery. | 30 days from the day of the surgery.
  Numbers of survivors will be assessed on 30th day after the surgery. The result will be displayed as a percentage of examined group.
Percentage of patients suffering from major cardiovascular event during 30 days after the surgery. | 30 days from the day of the surgery.
  Occurence of stroke or acute coronary syndrome will be assessed during period of 30 postoperative days. The result will be displayed as a percentage of examined group.
Percentage of patients suffering from postoperative delirium during 7 days after the surgery. | 7 days after the surgery.
  Occurence of postoperative delirium will be assessed during 7 days after the surgery. The result will be displayed as a percentage of examined group.

SECONDARY OUTCOMES:
Pain score after surgery | first 24 hours after surgery
  Patients will be asked about their pain ranks 6 and 24 hours after surgery. The NRS score will be used (0 to 10) where 0 is no pain and 10 is extremely severe pain.
Opioid consumption | first 24 hours after surgery
  Opioid (eg morphine) consumption will be noted

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No